CLINICAL TRIAL: NCT06863649
Title: Measuring Biomarkers for Health in Community Environments: eMBraCE Activity Program; Short Term Effect of Using Non-immersive Gamified Exercises on Chronic Shoulder Pain in People With Chronic Stroke.
Brief Title: Short-term Effect of Using Non-immersive Gamified Exercises on Chronic Pain in People With Stroke.
Status: Recruiting | Type: Observational
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: 22-05-04-B-02
Record Dates: First submitted 2025-01-20; First posted 2025-03-07 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Stroke Patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- chronic people with stroke
  Interventions: Other: Gamified NON-IMMERSIVE VIRTUAL REALITY EXERCISES; Other: video-based exercises

INTERVENTIONS:
Other: Gamified NON-IMMERSIVE VIRTUAL REALITY EXERCISES — The game phase lasts for 2 minutes. These targets are challenging for the participant.
Other: video-based exercises — The participant will exercise by replicating the exercises demonstrated in a 2-minute video, recorded with the same movement patterns that they will find in the gamified intervention.

SUMMARY:
Rehabilitation after stroke is essential to minimize permanent disability. Gamification of exercises has emerged as a promising strategy for increasing motivation and rehabilitation efficacy in people with stroke. However, there is a gap in understanding how exercise gamification can aid in pain management among people with stroke who are experiencing shoulder pain difficulties.

This study aims to evaluate the short-term effect of using gamified non-immersive exercises on shoulder pain level, upper limb range of motion, and shoulder and elbow muscle activities while doing different activities in people with chronic stroke. The study will be conducted using an observational study design. Various lab assessments include measuring the ROM of the shoulder (MOCAP), EMG, FNIRS, pain intensity using VAS scale, and muscles activities patterns across upper limb joints.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing motor difficulties in using the paretic arm, with some use of hand/arm as determined by therapist
* Not participating any other intervention studies
* Male/female ≥18 years old
* Had a stroke requiring with any degree of arm mobility.
* Capacity to consent to participate
* Able to communicate adequately in English with the research team
* Mild or moderate pain in shoulder or upper limb (below 6 and more than 2on the VAS scale).
* Able to walk without any assistant at least for ten meters

Exclusion Criteria:

* Any medical condition compromising the safety or the ability to take part to the study as determined by the therapist (such as insufficient vision or hearing, upper limb condition not linked to stroke, uncontrolled blood pressure, uncontrolled diabetes, co-morbidity)
* History of more than one epileptic seizures since stroke onset or uncontrolled epileptic seizure
* Unable to follow two stage command
* Moderate to severe hemi-spatial neglect compromising the ability to take part to the study, as determined by rehab team
* Severe spasticity (more than 2 on the modified Ashworth scale)
* Any device preventing use of EMG, FNIRS i.e. DBS or pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include 30 individuals of both genders experiencing shoulder pain. The inclusion criteria require participants to be over the age of 18, experiencing motor difficulties, have a stroke requiring upper/limb mobility rehabilitation, and be able to consent and communicate. Participants should not have other medical conditions that compromise the safety or ability to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Pain level | Pain levels will be measured on the same day, immediately before and immediately after the intervention.
  Pain levels will be measured using VAS (visual analog scale).
Range Of Motion | ROM will be measured immediately before starting the interventions
  This will be measured by doing Arm Abduction, Arm Flexion, Hand to Mouth, and Hand to Head. They will be measured by using a specific questionnaire of how well the participant can do each of them.
Brain Activity using fNIRS (Functional near-infrared spectroscopy) | Brain acticities will be measured when participants are asked to do the interventions. It means the time frame will be same as duration of the interventions, approximately 20 minutes.
Muscle activity using EMG (Electromyography) | Muscle activities will be measured when participants are asked to do the interventions and assessemnts. It means the time frame will be same as duration of the interventions and assessemnts, approximately one and half hours.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Dawes, Principal Investigator — University of Exeter; Maedeh Mansoubi, PhD, Principal Investigator — University of Exeter
Locations (1):
- Vsimulator, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No